CLINICAL TRIAL: NCT06460584
Title: Effect of Incentive Spirometer and Pursed Lip Breathing to Improve Dyspnea, Oxygen Saturation and Hospital Stay After Whipple Procedure.
Brief Title: Effect of Incentive Spirometer and Pursed Lip Breathing After Whipple Procedure.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0368
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hospital Stay
Keywords: Dyspnea,; Incentive Spirometer; Oxygen Saturation; Whipple procedure
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pursed Lip Breathing (Experimental): For the use of PLB exercise, the intervention will be given every day till the patient discharged from hospital. Patient will perform 5 sets. In each set, 10 times will be included
  Interventions: Other: Pursed Lip Breathing
- Incentive Spirometer (Active Comparator): The intervention will be given every day till the patient discharged from hospital. Patient will perform 5 sets, in each set, 10 times will be included and hold for 3 seconds but not more than 5 seconds. Reading will be taken on every 4rth POD and comparison will be done with 1st POD reading and so on.
  Interventions: Other: Incentive Spirometer

INTERVENTIONS:
Other: Pursed Lip Breathing — In each set, 10 times will be included. Reading will be taken from 1st POD and comparison will be done on each 4rth POD. Ask the patient to sit in a comfortable position and relax. Then, instruct the patient to take deep breath 12 through nose for two counts, and keep mouth closed. Inhale for 2 seconds. Now, ask the patient to purse the lips as if the patient was going to gently flicker the flame of candle. Now the patient will breathe out gently while counting for 4 seconds.
  Arms: Pursed Lip Breathing
Other: Incentive Spirometer — For the use of flow based IS, the Patient will be sited in a comfortable Position (Semi-Recumbent Position Of 45 Degrees), With a Pillow under the knees or Semi-Fowler Position on bed, and then asked to perform this technique with the same order to ensure that she / he understands the process. The patient will be instructed to inhale with a slow continuous and deep breathing, and hold for a period of not less than 5 seconds and exhale passively. And is instructed to hold the spirometry upright to perform slowly inhalation, thus lifting the ball. At the end of the evaluation of respiratory measures for patients with lung function, and then compare the results with the previous results. IS will be recommended to be performed by patient every 10 breaths hourly and 5 times per day.
  Arms: Incentive Spirometer

SUMMARY:
Whipple procedure is one of the most complex surgeries among hepatobiliary surgeries. It has named as Pancreaticoduodenectomy. It can cause many PPCs. Lung volumes are reduced due to atelectasis and pneumonia. Incentive spirometer (IS) is used to prevent PPCs. Due to general anesthesia, atelectasis is among most frequent PPCs. Pursed Lip Breathing (PLB) supports the patient to control the breath. The shriveling lips provide resistance to the air flowing out of the lungs. Airway collapse can be prevented by prolonged exhalation. Dyspnea occurs during 6MWT when patient performs walk in corridor. The aim of this study is to check the effect of Incentive Spirometer and Pursed Lip Breathing to improve dyspnea, oxygen saturation and hospital stay after Whipple procedure. This research of RCT will check the effect of IS and PLB by taking sample size of 60 post-operative patients through convenient sampling technique by allocating them randomly in group A and group B. Group A will receive PLB and group B will receive IS with baseline treatment chest percussions up to the duration of every day till discharge (reading will be collected on every 4rth day), dyspnea will be assessed through 6MWT and measured by Modified MRC dyspnea scale. The data will be analyzed through SPSS 26.

ELIGIBILITY:
Inclusion Criteria:

* Age (45 to 70)
* Type of Abdominal Surgery (Whipple Procedure) (11)
* Gender (Male and Female)
* Patients who has no history of pulmonary disease
* Smokers and nonsmokers

Exclusion Criteria:

* COPD (COPD patient with postoperative whipple procedure)
* Heart patient (patients who had history of heart disease along with whipple procedure)
* Uncontrolled Hypertension (patients who has have history of uncontrolled hypertension in postoperative whipple procedure)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Pulse Oximeter | baseline and fourth week
  Pulse oximetry is a simple and non-invasive method used to examine oxygen saturation (SpO2) in various parts of body. Convenient use, speed and high accuracy in detection of hypoxia and continuous monitoring of patients are other features of pulse oximetry
Modified MRC Dyspnea Scale | baseline and fourth week
  Medical Research Council (MRC) dyspnea scale the first clinical scale for the determination of dyspnea, is a 5-point scale based on the sensation of breathing difficulty experienced by the patient during daily life activities Patients, reading the 10 scale, are invited to recognize their own level of respiratory fatigue or, as is more often the case, the MRC can be directly administered
6-MWT | baseline and fourth week
  For the performance ability in many cardiopulmonary diseases, the most commonly used assessment tool is six minute walk test (6MWT). It has been widely used in research to evaluate the exercise capacity of various patient population (15). The test is standardized and reproducible self-paced exercise test. Patient is being asked to walk in a long hallway corridor for 6 minute between two cones on a flat surface. Ask the patient to keep walking. If the patient feels dyspnea, he or she may sit for a while. In healthy subjects with no history of pulmonary disease, the 6-min walk distance ranges from 400 to 700 m

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Afzal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zayed Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karim SAM, Abdulla KS, Abdulkarim QH, Rahim FH. The outcomes and complications of pancreaticoduodenectomy (Whipple procedure): Cross sectional study. Int J Surg. 2018 Apr;52:383-387. doi: 10.1016/j.ijsu.2018.01.041. Epub 2018 Feb 10. PMID 29438817
- [Background] Kotta PA, Ali JM. Incentive Spirometry for Prevention of Postoperative Pulmonary Complications After Thoracic Surgery. Respir Care. 2021 Feb;66(2):327-333. doi: 10.4187/respcare.07972. Epub 2020 Aug 25. PMID 32843511